CLINICAL TRIAL: NCT01856998
Title: Therapeutic Equivalence Study of Propofol Using Target-Controlled Infusion of Propofol 2% (20 mg/mL) MCT Fresenius Compared With Diprivan® 20 mg/mL (AstraZeneca) in Patients Undergoing Elective Surgery
Brief Title: Therapeutic Equivalence (TE) Study of Propofol 2% MCT Fresenius (MCT=Medium-Chain Triglycerides) Compared With Diprivan® in Patients Undergoing Elective Surgery
Acronym: PropofolTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROP-001-CP3; 2012-005701-43 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: General Anesthesia; Elective Surgery
Keywords: Therapeutic Equivalence; Propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diprivan® 20 mg/mL (AstraZeneca) (Active Comparator): Dosage form: lipid emulsion
  Dosage: Initial effect-site target concentration: 5 μg/mL, if necessary increased by 1 μg/mL every 60 seconds until LOER
  Frequency: continuously (will be adjusted to keep Bispectral Index (BIS) between 40 and 60, however maintenance target concentration can be increased if a patient needs a BIS <40 with regard to individual condition and the respective surgery)
  Duration: Until end of surgery
  Interventions: Drug: Diprivan
- Propofol 2% (20 mg/mL) MCT Fresenius (Experimental): Dosage form: lipid emulsion
  Dosage: Initial effect-site target concentration: 5 μg/mL, if necessary increased by 1 μg/mL every 60 seconds until LOER
  Frequency: continuously (will be adjusted to keep Bispectral Index (BIS) between 40 and 60, however maintenance target concentration can be increased if a patient needs a BIS <40 with regard to individual condition and the respective surgery)
  Duration: Until end of surgery
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol
  Arms: Propofol 2% (20 mg/mL) MCT Fresenius
Drug: Diprivan
  Arms: Diprivan® 20 mg/mL (AstraZeneca)

SUMMARY:
The purpose of this study is to evaluate the therapeutic equivalence, based on pharmacodynamic parameters of Propofol 2% (20 mg/mL) MCT Fresenius and Diprivan® 20 mg/mL (AstraZeneca), administered by target controlled infusion (TCI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years and <65 years old
2. Able to understand and give signed and dated written informed consent
3. Body mass index (BMI) ≥20 and ≤30 kg/m² at screening
4. ASA (American Society of Anesthesiologists) physical status 1 or 2
5. Undergoing elective, minor orthopedic, vascular, urological, or gynecological surgery
6. Patients should be affiliated to a social security scheme and benefit from the corresponding rights and cover

Exclusion Criteria:

1. The following planned procedures are to be excluded:

   * Day surgery
   * Emergency surgery
   * Total hip or total knee replacement
   * Requiring opening of the great cavities of the body (cranium, thorax, peritoneum, or pelvis)
   * With routine risk, even if low, of hemorrhage severe enough to require administration of colloid or blood products
   * With routine risk, even if low, of death during or soon after the procedure
   * Vascular surgery involving the aorta, venae cavae, iliac arteries, or femoral arteries
2. Intended administration of IV medications through a central venous catheter (Note: a central venous catheter may be used to obtain Pharmacokinetic (PK) samples, though only if no port of the catheter is being used for administration of any other product, including crystalloid infusion at more than a "keep line open" rate)
3. Administration of general anesthesia or propofol within the 7 days prior to randomization
4. History of hypersensitivity to propofol, eggs, soya, peanuts, or any other constituent of the study drugs
5. ASA physical status ≥3
6. History of major anesthesia complications including, but not limited to:

   * Clinically significant hypoxia
   * Profound hypotension
   * Anaphylaxis or anaphylactic reactions
   * Unpredictable anesthesia agent requirements
7. History of difficult airway management including, but not limited to:

   * Problematic artificial ventilation with face mask
   * Repeated difficulty of placement of laryngeal mask airway (LMA)
   * Difficult laryngeal intubation (Cormack-Lehane grade 3 to 4) and requiring alternative technique e.g. fibre-optic or awake laryngeal intubation
8. History of difficult venous access
9. Myocardial infarction within 6 months of randomization or a cardiac reperfusion procedure within 6 weeks of randomization
10. Significant respiratory, cardiovascular, liver or renal disease as assessed by investigator
11. Active systemic infection (localized infection related to surgical procedure is allowable as long as there is no indication of systemic involvement)
12. History of psychiatric disorder, including use of sedatives or antidepressants for any reason, within 6 months prior to randomization
13. Alcohol or other substance abuse within 2 years prior to randomization, as well as for the duration of the study
14. Use of medication that could reduce the subject's respiratory and/or cardiac output
15. Female subjects who are pregnant, breastfeeding, or lactating
16. Hemoglobin <7.5 g/dL at screening or randomization
17. Platelets <50,000 x 10³/μL at screening or randomization
18. ECG findings detected at screening not consistent with the subject's medical history or warranting cardiology review
19. Participation in an interventional clinical study within 6 months of screening
20. History of Propofol infusion syndrome

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Time to Loss of Eyelash Reflex (LOER) | Every ten seconds from the initiation of TCI anesthesia device until LOER occurs up to 150 seconds. If LOER has not occurred within this timeframe, target propofol concentration to be increased by 1 μg/mL every 60 seconds until LOER is observed.
  The overall timeframe until LOER is observed depends on the patient and varies from only a few seconds up to 240 seconds in total.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Sztark, Professor, Principal Investigator — CHU de Bordeaux, Groupe Hospitalier Pellegrin
Locations (1):
- CHU de Bordeaux, Groupe Hospitalier Pellegrin, Bordeaux, France